CLINICAL TRIAL: NCT06299462
Title: Efficacy Evaluation of Post-transplant Cyclophosphamide-based Graft-versus-host Disease Prophylaxis with ATG, Calcineurin Inhibitor-free, for Matched-sibling or Matched-unrelated Transplantation
Brief Title: PTCy and ATG for MSD and MUD Transplants
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTCy-ATG-001
Record Dates: First submitted 2023-03-13; First posted 2024-03-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: posttransplant cyclophosphamide; ATG; calcineurin-free GVHD prophylaxis; graft-versus-host disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patients with a matched sibling donor will be assigned to the PTCy+ATG4.l0 arm, while patients with a matched unrelated donor will be assigned to the PTCy+ATG5.0 arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matched-sibling donor transplants (Experimental): Matched sibling transplants will receive PTCy + ATG4.0
  Interventions: Drug: Cyclophosphamide injection; Drug: ATG 4.0
- Matched unrelated donor transplants (Experimental): Unrelated transplants will receive PTCy + ATG5.0
  Interventions: Drug: ATG 5.0; Drug: Cyclophosphamide injection

INTERVENTIONS:
Drug: ATG 5.0 — ATG 2.5 mg/kg on days -3 and -2
  Arms: Matched unrelated donor transplants
Drug: Cyclophosphamide injection — Cyclophosphamide 50 mg/kg on days +3 and +4
Drug: ATG 4.0 — ATG 2.5 mg/kg on day -2 + 1.5 mg/kg on day -3
  Arms: Matched-sibling donor transplants

SUMMARY:
Hematopoietic stem cell transplantation is a curative treatment for a number of benign and malignant hematologic diseases. One of the key parts of hematopoietic stem cell transplantation is the prophylaxis of graft-versus-host disease. Since the end of the 1970s, with the introduction of cyclosporine, calcineurin inhibitors (cyclosporine and tacrolimus) have become part of almost all prophylactic regimens, even though they are a group of drugs with a poor toxicity profile that requires monitoring. constant serum level. Since 2008, post-transplant cyclophosphamide has been introduced with great success, associated with a calcineurin inhibitor and mycophenolate, in the prophylaxis of graft-versus-host disease in haploidentical transplantation (50% matched).

Since then, in view of this enormous success, efforts have been made to incorporate post-transplant cyclophosphamide in matched related and unrelated transplants, or with a mismatch.

This is a prospective, 2-arm, non-randomized study. Arm 1, with related donors, and arm 2, with unrelated donors. Patients will be allocated in these arms according to donor availability (patients with a matched-sibling donor will receive a matched-sibling transplant; patients with no related donors but with unrelated donors, an unrelated transplant).

Patients who are ready for transplantation with matched-sibling or unrelated donors will be recruited to participate in the study.

The stem cell collection target will be 5E6 CD34/kg recipient weight for peripheral source. If a quantity greater than this is collected, the remainder will be cryopreserved according to the institutional protocol.

Graft-versus-host disease prophylaxis will be performed on D+3 and D+4 with cyclophosphamide and with ATG on D-3 and D-2 for matched-sibling or unrelated donors transplants.

ELIGIBILITY:
Inclusion Criteria:

* Patient with (1) acute leukemia in first or second remission; (2) myelodysplasia with less than 20% blasts; (3) Hodgkin's or non-Hodgkin's lymphoma, in partial remission after salvage therapy
* Who will receive a related or unrelated, HLA-compatible transplant;
* Who is a transplant candidate with FluMel, FluTBI, CyTBI, BuCy or BuFlu conditioning;
* Peripheral blood source;
* Age between 18 and 60 years.

Exclusion Criteria:

- Hepatic dysfunction (transaminases x2 the normal value)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of grades III-IV acute GVHD by the MAGIC criteria | 6 months
  Cumulative incidence of acute graft-versus-host disease, grades III-IV by the MAGIC criteria

SECONDARY OUTCOMES:
Cumulative incidence of grades II-IV acute GVHD by the MAGIC criteria | 6 months
  Cumulative incidence of acute graft-versus-host disease, grades II-IV by the MAGIC criteria
Cumulative incidence of steroid-refractory acute GVHD as defined by Mohty et al PMID 32756949 | 6 months
  Cumulative incidence of steroid-refractory graft-versus-host disease
Cumulative incidence of chronic GVHD as defined by the NIH criteria | 3 years
  Cumulative incidence of chronic graft-versus-host disease
Cumulative incidence of steroid-requiring chronic GVHD as defined by the NIH criteria | 3 years
  Cumulative incidence of steroid-requiring chronic graft versus host disease
Cumulative incidence of non-relapse mortality, i.e., death not following disease relapse | 3 years
  Cumulative incidence of death not caused by primary malignant disease or following relapse
Cumulative incidence of relapse, defined as > 5% blasts in bone marrow or 1% blasts in peripheral blood (acute leukemias/myelodysplasia) or biopsy proven relapse or positve PET-CT (lymphoma) | 3 years
  Cumulative incidence of relapse of primary malignant disease
Rate of overall survival | 3 years
  Death by any cause
Rate of disease-free survival (death or relapse) | 3 years
  Composite outcome of death or primary disease relapse
Cumulative incidence of clinically significant CMV reactivation (which led to antiviral treatment) | 3 year
  Incidence of cytomegalovirus reactivation
Cumulative incidence of posttransplant lymphoproliferative disorder (biopsy-proven or positive EBV PCR combined with clinical symptoms) | 3 years
  Incidence of posttransplant lymphoproliferative disorder
Cumulative incidence CMV disease (biopsy-proven CMV disease OR suggestive CMV+ BAL) | 3 years
  Cumulative incidence of cytomegalovirus disease
Measuremnt of quality of life using the FACT-BMT scale | 2 years
  Measurement quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo J Arcuri, MD, PhD, Principal Investigator — Instituto Nacional de Cancer
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Upon finalization of the study, data will be shared on reasonable requests.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code